CLINICAL TRIAL: NCT07368764
Title: The Suitability of Tience® for the Treatment of Acne Scars
Brief Title: The Suitability of Tience® for Treating Acne Scars
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Linio Biotech Oy (Industry)
Collaborators: Clinius Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT-009
Record Dates: First submitted 2026-01-20; First posted 2026-01-27 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Acne; Acne Scars
Keywords: acne scars; skin regeneration; skin regeneration treatment; substance of human origin; the healing of damaged skin; moderate, severe acne scars; skin diseases; Acne Vulgaris
MeSH Terms: conditions — Acne Vulgaris; Lymphoma, Follicular; Skin Diseases | interventions — Injections, Intradermal

STUDY DESIGN:
Intervention Model Description: Enrolled participants will be pseudorandomized to receive 3 Tience® Intradermal injection treatments to either the left or right facial half.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intradermal injections of Tience® cell-free allogeneic adipose tissue product (Experimental): Split face, Intradermal injections of Tience® cell-free allogeneic adipose tissue product on one side of the face.
  Interventions: Procedure: Intradermal injections

INTERVENTIONS:
Procedure: Intradermal injections — Three treatment sessions involving intradermal injections of the Tience cell-free allogeneic adipose tissue product administered to one side of the face.

SUMMARY:
This is an open-label, single-center, split-face, pseudo-randomized clinical trial designed to evaluate the efficacy and safety of a human-derived, cell-free adipose tissue derivative (Tience® ), for treating moderate to severe acne scars. Participants will receive three treatment sessions over a three-month period: on Day 0, Day 30, and Day 90. Treatment will be administered via injections to acne-scarred areas on one side of the face. The untreated side will be treated after the follow-up period. Outcomes will be evaluated over a twelve-month period using investigator clinical assessments, patient self-evaluation and VISIA skin analysis system to monitor changes in scar severity and overall skin quality.

DETAILED DESCRIPTION:
Tience®, a human adipose tissue derivative, is intended to be used in the human body for its original purpose to supplement and replace local extracellular matrix deficiencies in soft tissue, including skin. Tience provides a temporary conductive environment into the injured area. This facilitates the ability of local cells to re-populate the damaged soft tissue and skin area, thereby enabling the deposition of extracellular matrix and repair of the tissue. Tience is authorized for treatment of wounds, scars and soft tissue defects.

The purpose of this study is to determine whether the product is suitable for the treatment of acne scars, and to collect safety data on the use of Tience® in this indication.

ELIGIBILITY:
Inclusion Criteria: healthy volunteers aged 18-40 years who have at least 3-year- old acne scars on their cheeks.

-

Exclusion Criteria:

* pregnancy or nursing
* cancer or ongoing cancer treatment
* an active skin disease
* Fitzpatric scale 4-6 skin type
* a strong medication used for treating severe acne (e.g., Isotretinoin)
* active acne or Herpes
* antihistamine medication (if the medication can be paused for 7 days during study visits, participation is possible)
* use of biological medications
* tendency for excessive scar formation
* tendency for urticaria (hives)
* systemic medication affecting immunity
* autoimmune disease
* known disease affecting blood clotting (bleeding or thrombosis tendency) (e.g., von Willebrand disease)
* are allergic to the product being studied or any of its ingredients
* smoke

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-05-01 (Actual); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Postacne Scarring: A Qualitative Global Scarring Grading System (Goodman and Baron) | Participants are evaluated at four time points: Day 0 (prior to the first treatment), Day 30 (prior to the second treatment), Day 90 (prior to the third treatment), and Day 180 (final evaluation visit)
  The researcher will grade the participants' acne scars before treatments, and at final evaluation visit using the Goodman and Baron qualitative and quantitative acne scar scales.
  For the Goodman and Baron quantitative scar scale, scars will be categorized according to morphology by recording the number of mild, moderate, severe, and hypertrophic lesions. A total score (range: 0-84), with higher scores indicating greater severity and number of scars.
  For the Goodman and Baron qualitative scar scale, scars will be classified into four categories: Grade 1= macular, Grade 2= mild, Grade 3= moderate, and Grade 4= severe.
Visia® Gen7 Skin Analysis System | Before first treatment, Day 30 before second treatment, Day 90 before third treatment, and Day 180 evaluation visit.
  A Visia Gen7 skin analysis will be performed on the study participants before each treatment and at final evaluation visit 180 days after first treatment.
Self assessment of study participants | 180 days
  Subjective self-assessment of acne scars by study participants before each treatment and at the final evaluation visit.

SECONDARY OUTCOMES:
The adverse reactions and adverse events assessment questionnaire for the participants | Assessment will be conducted 7 days after each treatment.
  The questionnaire for the study participants of the side effects 7 days after each treatment. Parameters: itching, edema, bruising, tingling, pinpoint bleeding, erythema, needle marks, injection site pain, allergic reaction, skin tenderness, dizziness or feeling unwell during the treatment. The evaluation is conducted using a scale from 0 to 10, where 0 indicates no symptoms and 10 indicates the most severe possible symptoms, along with the duration of the symptoms.
Descriptive safety evaluation of the researcher including incidence rates of adverse events | 180 days
  All adverse events related to study product or its administration, incidence of AEs, withdrawals due to AEs and all Serious Adverse Events (SAEs) will be assessed. All adverse events will be reported and followed until resolved.
The adverse reactions and events assessment questionnaire for the researcher | Day 0 the first treatment, Day 30 the second treatment, and Day 90 the third treatment.
  The questionnaire for the researcher of the side effects after each treatment. Parameters: edema, bruising, pinpoint bleeding, erythema, injection site pain, allergic reaction. The evaluation is conducted using a scale from 0 to 10, where 0 indicates no symptoms and 10 indicates the most severe possible symptoms of the study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Laura Bouchard, MD, PhD, Principal Investigator — Aava Kamppi Medical Centre
Locations (1):
- Aava Kamppi Medical Centre, Helsinki, Finland

IPD SHARING:
Plan to Share IPD: No